CLINICAL TRIAL: NCT07052149
Title: Cervical Muscle Stabilization Versus Neck Proprioception Training on Neck Flexors Endurance in Adolescents With Forward Head Posture
Brief Title: Stabilization vs Proprioception Training on Neck Flexor Endurance in Adolescents With Forward Head Posture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, walaa eldesoukey heneidy, Lecturer of Physical Therapy, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Forward Head Posture
Record Dates: First submitted 2025-06-19; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Forward Head Posture

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical muscle stabilization (Experimental): 15 adolescent with foreward head posture receiving Cervical muscle stabilization exercises
  Interventions: Other: cervical muscle stabilization exercises
- Proprioceptive training (Experimental): 15 adolescent with foreward head posture receiving Proprioceptive training
  Interventions: Other: Proprioceptive training

INTERVENTIONS:
Other: cervical muscle stabilization exercises — deep cervical muscle stabilization exercises, 15 minutes, 3 sessions per week for two months
  Arms: Cervical muscle stabilization
Other: Proprioceptive training — proprioceptive training, 15 minutes, 3 sessions per week for two months
  Arms: Proprioceptive training

SUMMARY:
Forward Head Posture (FHP) is a common postural deviation among adolescents, often resulting from prolonged screen use and poor ergonomic habits. It is characterized by an anterior positioning of the head relative to the vertical midline of the body, leading to altered cervical spine mechanics and muscle imbalances. One of the key consequences of FHP is the reduced endurance of deep neck flexor muscles, which play a crucial role in cervical stability and postural control.

Cervical muscle stabilization exercises and proprioceptive training are two widely used interventions aimed at improving neuromuscular control and endurance of cervical muscles. While both methods have shown benefits in postural correction, their relative effectiveness in enhancing neck flexor endurance in adolescents with FHP remains unclear.

This study aims to compare the effects of cervical muscle stabilization versus neck proprioception training on the endurance of deep neck flexors in adolescents with Forward Head Posture.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent with forward head posture
* Their age ranged from 16 to 18 years
* They had normal height, weight, and BMI (BMI percentile ≥5 and <85) relative to their age.
* They were free from any medical condition or musculoskeletal deformity that could affect posture or interfere with the assessment or intervention procedures
* They were free from any visual or hearing problem

Exclusion Criteria:

* • Athletic adolescent

  * Adolescent with congenital or acquired spinal deformities
  * Adolescent having any Injury to the neck or upper extremity and history of joint inflammation
  * Adolescent with neurological, musculoskeletal and cardiopulmonary disease that limit their movement
  * Adolescent with cognitive disorders, or vision disorders not corrected by glasses

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
cranio vertebral angle | pretreatment and after 2 months of intervention
  meauring craniovertebral angle using kineovia software

CONTACTS AND LOCATIONS:
Overall Officials: Hala I Kassem, Professor, Study Chair — Professor
Locations (1):
- Walaa HENEDY, Damietta, Damietta Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No